CLINICAL TRIAL: NCT03623412
Title: Women With Minor Degrees of Glucose Intolerance and the Postpartum Glucose
Brief Title: Women With Minor Degrees of Glucose Intolerance and the Postpartum Glucose Tolerance Test
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Clalit Health Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 0068-18
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Glucose Tolerance Impaired in Pregnancy
MeSH Terms: interventions — Glucose Tolerance Test

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One abnormal value (Experimental): Women with only one abnormal value on OGTT (Oral Glucose Tolerance Test) during pregnancy
  Interventions: Diagnostic Test: 75g oral glucose tolerance test
- GDM (Active Comparator): Women with two abnormal values on OGTT during pregnancy - diagnosis=GDM
  Interventions: Diagnostic Test: 75g GTT

INTERVENTIONS:
Diagnostic Test: 75g oral glucose tolerance test — Women with one abnormal value in the OGTT during pregnancy (minor degree of glucose intolerance) will be offered a post-partum 75g GTT (Glucose Tolerance Test), similar to that offered to women with GDM
  Arms: One abnormal value
Diagnostic Test: 75g GTT — post-partum GTT
  Arms: GDM

SUMMARY:
The aim of this study is to offer a 75g postpartum glucose tolerance test to women with minor degrees of glucose intolerance and to assess if these women are significantly different from women who were diagnosed as GDM (Gestational Diabetes Mellitus)

ELIGIBILITY:
Inclusion Criteria:

* healthy women (without pre-existing diabetes) who underwent an OGTT during pregnancy

Exclusion Criteria:

* pre-existing diabetes, or failed to perform the OGTT

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-08-15 (Estimated); Primary Completion 2019-09-15 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Positive post-partum GTT results | 6-12 weeks post partum